CLINICAL TRIAL: NCT01719042
Title: Improving Tolerance of Treatment of Pulmonary Mycobacterium Avium Complex Infections
Brief Title: Improving Tolerance of Treatment of Pulmonary MAC Infections
Acronym: ITT-MAC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No recruitment was achievable
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 187-2012
Record Dates: First submitted 2012-10-22; First posted 2012-11-01 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Mycobacterium Avium Complex; Adverse Effects
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection | interventions — Ondansetron; Ensure Plus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zofran (8mg) (Active Comparator): Participant will take Zofran (8mg) once per day before taking their antibiotic regimen
  Interventions: Drug: Zofran (8mg)
- Ensure (Active Comparator): Subject will drink a can of Ensure before taking their antibiotic regimen
  Interventions: Dietary Supplement: Ensure

INTERVENTIONS:
Drug: Zofran (8mg) — Subject will take 8mg of Zofran before taking antibiotic regimen and will record symptoms in a diary just before taking medication and two hours after taking medication every day for two weeks
  Other Names: Ondansetron
  Arms: Zofran (8mg)
Dietary Supplement: Ensure — Subject will drink one cam of Ensure before taking antibiotic regimen and will record symptoms in a diary just before taking medication and two hours after taking medication every day for two weeks
  Other Names: Ensure Plus
  Arms: Ensure

SUMMARY:
The purpose of this study is to improve tolerance of treatment of pulmonary Mycobacterium avium Complex disease via the use of therapeutic drug monitoring and the addition of anti-nausea medication or dietary supplements to the patients' daily drug regimen. The aims of this study are to use (1) Zofran® (Ondansetron 8mg), an anti-nausea medication or (2) a dietary supplement to decrease medication related gastrointestinal side effects of medications used to treat Mycobacterium avium Complex.

DETAILED DESCRIPTION:
As part of this study, investigators will review medical records to be sure that the patient meets the required criteria and is healthy enough to take part in this study.

The study will consist of five separate visits to the Clinical research Center at the University of Florida and each visit will last anywhere from 6-8 hours. Patients will be given a diary of questionnaires where they will record when they take their medication and any side effects they might have. Patients will also have Electrocardiograms (ECGs) to make sure they are healthy enough to be a participant in the study and to measure the effects of their medication on their heart. During this study, patients will continue treatment of their Mycobacterium avium Complex infections. Patients will be observed taking their medication on each of the five separate days. On each of these days patients will have blood drawn at 2 and 6 hours after their drugs are taken in order to measure drug levels in their blood. We will also use this blood to measure levels of proteins and hormones and to make sure the medications are not affecting the patient's heart. The patient will fill out several questionnaires and do a dietary assessment online. Investigators will assess the patient's body make-up using a device called the Bod Pod. The patient will also be assigned to one of two treatment groups: (1) Ondansetron 8mg (Zofran®, GlaxoSmithKline, Research Triangle Park, NC) every morning before breakfast versus (2) a dietary supplement prior to taking daily medication. The patient will be assigned to the first treatment group for a period of two weeks. On the third study visit investigators will switch the patient to the second group.

Although the incidence of tuberculosis has decreased in the United States over the last few decades, the incidence of chronic pulmonary infections with nontuberculous mycobacteria (NTM) appears to be increasing. Unfortunately, a common problem in the management of these infections is the inability of elderly patients to tolerate the currently recommended multidrug regimen of (1) azithromycin or clarithromycin, (2) rifampin or rifabutin, and (3) ethambutol. The most frequent adverse reactions of MAC treatment are gastrointestinal (GI), most commonly associated with the macrolides and rifampin. Although macrolide toxicity is generally dose-related, the role of routine monitoring of drug concentrations and subsequent dose adjustment has not been studied. The role of anti-emetics or dietary supplements to mitigate these symptoms is also not defined.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of Mycobacterium avium Complex with nodular bronchiectasis
* On daily treatment for Mycobacterium avium Complex consisting of 250mg of Azithromycin, 600mg of Rifampin, and 15mg/kg of Ethambutol
* Experiencing gastrointestinal symptoms due to their multi-drug treatment regimen
* Has access to the internet

Exclusion Criteria:

* Claustrophobia
* Currently smokes cigarettes
* Persons with disseminated Mycobacterium avium Complex infections
* Persons with a known and diagnosed immunosuppressive disorder (i.e. cancer, HIV)
* Persons with physician diagnosed Irritable Bowel Syndrome, Crohn's Disease, or Ulcerative Colitis
* Persons with moderate to severe kidney or liver dysfunction
* Persons who are co-colonized with an NTM aside from Mycobacterium avium Complex
* Persons who initially present with a prolonged QT interval (defined as greater 500 milliseconds) on any baseline ECG
* Previous adverse reaction or allergy to Zofran (Ondansetron)

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in Gastroparesis Cardinal Symptom Index Score | Change from baseline at the end of nine weeks
  A survey instrument used to assess the severity of patient-reported gastrointestinal symptoms in clinical trials

SECONDARY OUTCOMES:
Leptin | Baseline
  Leptin is a natural hormone produced by your body's fat cells and acts as a signal which tells your brain you are no longer hungry

OTHER OUTCOMES:
Change in QTc on Electrocardiogram greater than 500 milliseconds | Change from baseline at the end of nine weeks
  To determine if the drug-drug interaction of azithromycin and Zofran (ondansetron) causes significant prolongation of the corrected QT (QTc) interval in this population of older female patients

CONTACTS AND LOCATIONS:
Overall Officials: Kevin P Fennelly, MD, MPH, Principal Investigator — University of Florida